CLINICAL TRIAL: NCT04136262
Title: Tripterygium Wilfordii Hook F and Methotrexate for Postmenopausal Women With Rheumatoid Arthritis: a Randomized Controlled Trial
Brief Title: Tripterygium Wilfordii Hook F and Methotrexate for Postmenopausal Women With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, Guang'anmen Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018YFC1705204
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; Tripterygium wilfordii Hook F; methotrexate; postmenopausal women; randomized controlled trial
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tripterygium wilfordii Hook F (TwHF) plus methotrexate (MTX) (Experimental): Oral Tripterygium wilfordii Hook F 20mg thrice daily for 24 weeks. Oral methotrexate 10 mg per week for 24 weeks.
  Interventions: Drug: Tripterygium wilfordii Hook F (TwHF); Drug: Methotrexate
- TwHF (dummy) plus MTX (Placebo Comparator): Oral dummy Tripterygium wilfordii Hook F 20mg thrice daily for 24 weeks. Oral methotrexate 10 mg per week for 24 weeks.
  Interventions: Drug: Methotrexate; Other: Dummy Tripterygium wilfordii Hook F (TwHF)

INTERVENTIONS:
Drug: Tripterygium wilfordii Hook F (TwHF) — Oral Tripterygium wilfordii Hook F 20mg thrice daily for 24 weeks.
  Other Names: DND Pharm
  Arms: Tripterygium wilfordii Hook F (TwHF) plus methotrexate (MTX)
Drug: Methotrexate — Oral methotrexate 10 mg per week for 24 weeks.
  Other Names: XINYI Pharm
Other: Dummy Tripterygium wilfordii Hook F (TwHF) — Oral dummy Tripterygium wilfordii Hook F 20mg thrice daily for 24 weeks.
  Arms: TwHF (dummy) plus MTX

SUMMARY:
This study is a multicenter, randomized, double-blinded, controlled trial with two parallel arms. The aim of the study is to evaluate whether Tripterygium wilfordii Hook F combined with methotrexate (MTX) might be better than MTX alone for postmenopausal women with active rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
To compare the efficacy and safety of Tripterygium wilfordii Hook F (TwHF) and methotrexate (MTX) for postmenopausal women with active rheumatoid arthritis (RA), a multicenter, randomized controlled trial will be conducted. Three hundred postmenopausal women with active RA will be randomly allocated (1:1) to treatment with TwHF 20mg thrice daily and MTX 10 mg once a week for 24 weeks, or MTX plus dummy TwHF. The primary outcome is the percentage of participants with American College of Rheumatology 20% at week 24.

ELIGIBILITY:
Inclusion Criteria:

1. postmenopausal women, postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy;
2. diagnosed with RA as determined by meeting the 2010 ACR/EULAR classification criteria and having had RA for at least 6 weeks;
3. active disease at the time of enrollment as indicated by 28-joint Disease Activity Score (DAS28) greater than 3.2;
4. no prior exposure to oral glucocorticoids at a daily dose greater than 10 mg or to any biologic agents.

Exclusion Criteria:

1. RA combined with other autoimmune disease, such as adjuvant arthritis, lupus arthritis, or osteoarthritis;
2. RA combined with abnormal liver and kidney function;
3. severe chronic or acute disease interfering with attendance for therapy;
4. patients who had received DMARDs or biological therapy within one months before participating in this study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of ACR20 | week 24
  Percentage of Participants With American College of Rheumatology 20% (ACR20)

SECONDARY OUTCOMES:
Percentage of ACR50 | week 24
  Percentage of Participants With American College of Rheumatology 50% (ACR 50)
Percentage of ACR70 | week 24
  Percentage of Participants With American College of Rheumatology 70% (ACR 70)
RAMRIS score | week 24
  To explore the structural efficacy of Tripterygium wilfordii Hook F (TwHF) on synovitis, osteitis, and joint erosions as measured by MRI in postmenopausal women with active RA using the change in the RAMRIS score from Baseline to Week 24.
Mean 24-week Change in Disease Activity Score Based on 28-Joint Count (DAS28) | week 24
  Average difference between 24-week and Baseline DAS28
Change From Baseline in Modified Total Sharp X-Ray Score at Week 24 | week 24
  Modified Total Sharp Score (mTSS) is a measure of joint health, used in evaluation of inhibition of radiographic progression of disease
Patient Reported Outcomes (PRO) | week 24
  Patient-Reported Outcomes Scale

CONTACTS AND LOCATIONS:
Overall Officials: Quan Jiang, M.D, Principal Investigator — Guang' anmen hospital
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, China